CLINICAL TRIAL: NCT05542680
Title: Study on the Design and Application of Special Semi Recumbent Cushion for Postoperative Patients With Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCC2021C-266
Record Dates: First submitted 2022-08-28; First posted 2022-09-15 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Denture Liners

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): In the intervention group, the special cushion for semi recumbent position was used
  Interventions: Device: cushion
- Group 2 (No Intervention): Routine nursing intervention

INTERVENTIONS:
Device: cushion — In the intervention group, the special cushion for semi recumbent position was used
  Arms: Group 1

SUMMARY:
1. transform and produce the authorized utility model invention patent "a special cushion for semi recumbent position".
2. to verify the effect of using special semi recumbent cushion for postoperative patients with esophageal cancer.

DETAILED DESCRIPTION:
1. Make application-oriented achievement transformation products to provide new special semi recumbent auxiliary tools for patients with esophageal cancer after operation. Summarize the clinical experience and evidence, sign the project cooperation intention agreement with the manufacturer with production qualification, connect with the professional designer of the manufacturer and refine and improve the design scheme; The angle range, materials, fabrics and connection methods of the semi reclining cushion are closely combined with the clinical treatment and patient needs to meet the effectiveness, comfort and practicality of the patient's application; To produce semi reclining cushion products to provide semi reclining cushion for patients after esophageal cancer surgery that can be adjusted from multiple angles and take into account the skin protection function, which is conducive to preventing and alleviating reflux symptoms, improving the quality of life and reducing the risk of skin stress injury.
2. Implement and evaluate the effectiveness of the special semi reclining cushion after esophageal cancer surgery, apply the product to patients after esophageal cancer surgery, and evaluate the effect.

ELIGIBILITY:
Inclusion criteria:

1. transform and produce the authorized utility model invention patent "a special cushion for semi recumbent position".
2. to verify the effect of using special semi recumbent cushion for postoperative patients with esophageal cancer. 1. patients with pathologically confirmed esophageal cancer who underwent thoracoscopic resection and neck anastomosis;

2. age ≥ 18 years old; 3. able to read and fill in the questionnaire independently.

Exclusion criteria:

1. cognitive impairment or mental illness;
2. complicated with other serious diseases;
3. unwilling to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Reflux symptoms | 1 to 30 days after surgery
  Reflux Diagnostic Questionnaire RDQ The Reflux Diagnostic Questionnaire includes four symptoms: heartburn, acid reflux, regurgitation, and pain behind the sternum. The frequency and severity of symptoms range from 0 to 5 points. The highest score for symptom frequency and severity is 40 points. A higher score indicates more severe reflux, and a score exceeding 12 points indicates a preliminary diagnosis of gastroesophageal reflux disease

SECONDARY OUTCOMES:
Postoperative quality of life QLQ-C30 | 7 days after surgery
  European Organization for Research and Treatment of Cancer (EORTC): Quality of Life Questionnaire: EORTC QLQ-C30
  The Quality of Life Questionnaire QLQ-C30 is a tool for assessing the quality of life of cancer patients, with 30 items divided into 15 domains. The scoring method is as follows:
  For items 29 and 30, score from 1 to 7 according to the answer options; for other items, score from 1 to 4 according to the answer options .
  Add up the scores of the items included in each domain and divide by the number of items included, to get the raw score of that domain .
  Use the range method to perform a linear transformation, converting the raw score into a standardized score between 0 and 100 .
  For functional domains and overall health status/quality of life domain, the higher the score, the better the functional status and quality of life; for symptom domains, the higher the score, the more symptoms or problems (the lower the quality of life) .
Postoperative quality of life QLQ-OES18 | 7 days after surgery
  European Organization for Research and Treatment of Cancer (EORTC): Esophagus-specific QOL questionnaire: EORTC QLQ-OES18
  QLQ-OES18 is a module for assessing the quality of life of patients with esophageal cancer, which needs to be used together with the QLQ-C30 core questionnaire, with 18 items divided into 10 domains. The scoring method is as follows:
  For all items, score from 1 to 4 according to the answer options . Add up the scores of the items included in each domain and divide by the number of items included, to get the raw score of that domain .
  Use the range method to perform a linear transformation, converting the raw score into a standardized score between 0 and 100 .
  For functional domains and overall health status/quality of life domain, the higher the score, the better the functional status and quality of life; for symptom domains, the higher the score, the more symptoms or problems (the lower the quality of life) .
Skin pressure injury | 7 to 180 days after surgery
  The staging standard of pressure injury published by the national pressure sore Advisory Committee of the United States was applied to skin pressure injury

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No